CLINICAL TRIAL: NCT00427648
Title: Intravesical Alkalized Lidocaine for the Treatment of Overactive Bladder (OAB), a Randomized, Double-blinded Controlled Trial
Brief Title: Local Anesthetic Treatments for Overactive Bladder
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: funding ran out, poor accrual.
Sponsor: Frank Tu (Other)
Collaborators: Berlex Foundation (Other)
Responsible Party: Sponsor-Investigator, Frank Tu, Division Director, Gynecological Pain and Minimally Invasive Surgery, Department of Obstetrics and Gynecology, Endeavor Health
Organization: Endeavor Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH 06-092
Record Dates: First submitted 2007-01-26; First posted 2007-01-29 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Overactive Bladder
Keywords: Administration, Intravesical; Anesthetics, Local
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): xylocaine
  Interventions: Drug: alkalinized xylocaine
- 2 (Placebo Comparator): normal saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alkalinized xylocaine — 30 cc of 1% xylocaine and 10 cc of 0.9% sodium bicarbonate, dosed twice a week for three weeks
  Arms: 1
Drug: placebo — normal saline
  Other Names: normal saline
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether alkalized lidocaine instilled into the bladder is effective in the treatment of overactive bladder (OAB).

DETAILED DESCRIPTION:
Existing first-line treatments for overactive bladder are limited by requirements for chronic dosing and associated systemic side effects. Small case series suggest that bladder instillation of lidocaine may be effective in downregulating the afferent neuronal activity of a sensitized bladder, leading to elevation of the urge sensory threshold and decreasing detrusor activity. However, neither the effectiveness over placebo nor the durability of the response has been previously investigated.

Comparison(s): We propose a randomized, prospective double-blinded controlled trial to determine if a three-week trial of intravesical alkalized lidocaine instillation decreases symptoms of overactive bladder more than instillation of normal saline using a validated outcome instrument, the OAB-q.

ELIGIBILITY:
Inclusion criteria:

* Female patient, 18 years of age and older
* Overactive bladder defined as:

  * Urinary frequency defined as eight or more voids in a 24 hour period > 50% of days of the week
  * Symptoms of urgency
  * Symptoms of at least three months duration

Exclusion criteria:

* Positive urine culture in the past month, or more than 3 episodes of bladder infection in the last 2 months
* Stress or overflow urinary incontinence (determined by clinician) if more than 14 episodes of urinary incontinence per week; also insensate incontinence
* Pregnancy
* Seizure disorder or clinically significant renal disease, allergy to lidocaine, uninvestigated hematuria, or history of urinary/reproductive tract malignancy
* Post-void residual more than 200 cc

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank F. Tu, MD, MPH, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - NorthShore University HealthSystem, Evanston, Illinois
  - NorthShore University HealthSystem, Park City, Illinois

REFERENCES:
- [Background] Wein AJ, Rovner ES. Definition and epidemiology of overactive bladder. Urology. 2002 Nov;60(5 Suppl 1):7-12; discussion 12. doi: 10.1016/s0090-4295(02)01784-3. PMID 12493342
- [Background] HAINES JS, GRABSTALD H. Xylocaine; a new topical anesthetic in urology. J Urol. 1949 Dec;62(6):901. doi: 10.1016/S0022-5347(17)69020-7. No abstract available. PMID 15394388
- [Background] Parsons CL. Successful downregulation of bladder sensory nerves with combination of heparin and alkalinized lidocaine in patients with interstitial cystitis. Urology. 2005 Jan;65(1):45-8. doi: 10.1016/j.urology.2004.08.056. PMID 15667861
- [Background] Coyne K, Revicki D, Hunt T, Corey R, Stewart W, Bentkover J, Kurth H, Abrams P. Psychometric validation of an overactive bladder symptom and health-related quality of life questionnaire: the OAB-q. Qual Life Res. 2002 Sep;11(6):563-74. doi: 10.1023/a:1016370925601. PMID 12206577
- See also: Click here for more information about this study: Intravesical alkalized lidocaine for the treatment of overactive bladder (OAB), a randomized, prospective double-blinded controlled trial — http://www.northshore.org/clinicalservices/womenshealth/research/default.aspx?id=4429

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two medical clinic sites were used between January 2007 and March 2011, initially the Evanston Continence Center (Evanston, IL), and subsequently to augment recruitment, North Shore Urogynecology (Lake Forest, IL, added July 2009).
Pre-assignment Details: no wash out, no run-in
Groups:
- 1/Active: alkalinized xylocaine: 30 cc of 1% xylocaine and 10 cc of 0.9% sodium bicarbonate
- 2/Placebo: normal saline
Period: Overall Study
Arm/Group | 1/Active | 2/Placebo
Started | 12 | 10
Completed | 11 | 7
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Active | 2/Placebo | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: did not analyze patients eliminated from study due to protocol deviation and withdrawal due to AE
  years
    number analyzed (Participants) | 11 | 7 | 18
    (all) | 50.4 (11.3) | 54.3 (18.3) | 51.9 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 3 withdrawal of consents, and 1 patient with AE excluded from analysis
  Participants
    number analyzed (Participants) | 11 | 7 | 18
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 8 | 7 | 15
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22
length of OAB symptoms [Mean (Standard Deviation); unit: years] — Population: protocol withdrawals = 3 and 1 with AE not included
  years
    number analyzed (Participants) | 11 | 7 | 18
    (all) | 6.8 (10.2) | 7.7 (5.4) | 7.2 (8.5)
prior anticholinergic use [Count of Participants; unit: Participants] — Population: 3 withdrawals and 1 AE not included
  Participants
    number analyzed (Participants) | 11 | 7 | 18
    (all) | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Daily Voiding Episodes (by 3-day Voiding Diary) at Six Weeks.
Time Frame: 6 weeks
Population: only 16 participants completed this diary
Measure: Median (Inter-Quartile Range); unit: voids/day
Arm/Group | 1/Active | 2/Placebo
Number analyzed (Participants) | 10 | 6
voids/day | 9.5 [6.5 to 12.5] | 9 [6.75 to 9.75]
Statistical Analysis 1: Comparison: 1/Active vs 2/Placebo; null hypothesis - no difference in average number of voids between the 2 groups, power calculation estimated 40 participants needed per arm to show a 2 void difference between lidocaine and saline placebo; Test type: Superiority; p = 0.588, Kruskal-Wallis

2. Secondary Outcome: Median Number of Daily Voiding Episodes at 12 Months.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: voids/day
Groups:
- 1/Xylocaine: alkalinized xylocaine: 30 cc of 1% xylocaine and 10 cc of 0.9% sodium bicarbonate, dosed twice a week for three weeks
- 2/Normal Saline: placebo: normal saline
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 7 | 6
voids/day | 7 [7 to 9] | 8 [7.25 to 9.5]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.617, Kruskal-Wallis

3. Secondary Outcome: SF-12 Physical at 6 Weeks
Description: SF-12 physical is an abbreviated version of the SF-36 a widely used, general health care quality of life instrument. Scores range from 0-100, and higher scores are better outcomes.
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on scale
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 11 | 7
score on scale | 49 [39 to 56] | 56 [41 to 58]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.441, Kruskal-Wallis

4. Secondary Outcome: OAB-q (Symptom Scale) at 6 Weeks
Description: OAB-q SS is a 7 item overactive bladder symptom bother sub scale, ranging from 0-100, higher scores mean worse outcome for bother
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 11 | 7
score on a scale | 15 [11 to 36] | 28 [19 to 45]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.189, Kruskal-Wallis

5. Secondary Outcome: Global Assessment of Change - Frequency at 6 Weeks
Description: This is patient overall assessment of change in overactive bladder symptoms after treatment. 0% is no change, 100% is total resolution of symptoms
Time Frame: 6 weeks
Measure: Median (Inter-Quartile Range); unit: percent improvement
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 11 | 7
percent improvement | 40 [0 to 75] | 10 [5 to 27]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.342, Kruskal-Wallis

6. Secondary Outcome: Average Weekly NRS for Frequency at 6 Weeks
Description: NRS - numerical rating scale, 0-10 is the range, and higher scores are worse frequency
Time Frame: 6 weeks
Population: Not all women completed this measure
Measure: Median (Inter-Quartile Range); unit: score on a 0-10 scale
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 11 | 6
score on a 0-10 scale | 4 [3 to 6] | 4 [3 to 7]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.802, Kruskal-Wallis

7. Secondary Outcome: Cystometric Assessment of Maximal Bladder Capacity at 6 Weeks Only.
Description: This is based on retrograde infusion of sterile water into the bladder using a catheter, the maximum tolerated volume serving to define how much distension a woman can tolerate.
Time Frame: 6 weeks
Population: Not all women were able to return for cystometry
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | 1/Xylocaine | 2/Normal Saline
Number analyzed (Participants) | 8 | 6
mL | 316 [250 to 488] | 275 [200 to 325]
Statistical Analysis 1: Comparison: 1/Xylocaine vs 2/Normal Saline; Test type: Superiority; p = 0.366, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse event inventories were completed at each of 6 biweekly instillation visits and also at week 6, and 3,6, and 12 month followup visits
Arm/Group | 1/Active | 2/Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 3/11 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Active (N=11) | 2/Placebo (N=7)
bladder infection (Renal and urinary disorders) | 3 (3) | 2 (2)
pain in lower abdomen (General disorders) | 1 (1) | 0 (0) — week 3 only
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — week 3 only
pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
dysuria (Renal and urinary disorders) | 1 (1) | 2 (2)
urinary hesitancy (Renal and urinary disorders) | 1 (1) | 0 (0)
light headedness (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 0 (0)
sleepiness (General disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include the large amount of women unwilling to participate, the repeated need for catheterization for six instillations and two cystometries, the loss of subjects to follow-up, and some missing diaries of recorded daily voids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No